CLINICAL TRIAL: NCT00972452
Title: Acute Cardiovascular and Metabolic Effects of Exercise Training in Individuals
Brief Title: Blood Flow Responses to an Oral Glucose Tolerance Test in Type 2 Diabetes
Acronym: OGTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MUIRB1135317
Record Dates: First submitted 2009-09-04; First posted 2009-09-07 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Type 2 Diabetes; Insulin Resistance
Keywords: Type II Diabetes; Insulin Resistance; Exercise; Continuous Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise (Experimental): 5-10d exercise training
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — short period of exercise training (5-10 days)

SUMMARY:
The investigators wish to determine whether a short period of exercise training (5-10 days) improves the metabolic and cardiovascular response of people with or at risk of developing type 2 diabetes to eating a meal. In healthy people, blood flow to skeletal muscles increases after eating a meal, and this helps to regulate blood sugar levels by delivering blood sugar to muscles where it can be stored or metabolized. In people with or at risk of type 2 diabetes, blood flow does not increase as much after eating a meal, and this may contribute to elevated blood sugar concentrations observed in these individuals. The investigators wish to determine whether exercise can improve this response.

DETAILED DESCRIPTION:
Insulin resistance is characterized by decreased sensitivity to the metabolic actions of insulin (glucose disposal) and is a hallmark of obesity and type 2 diabetes (T2D). Insulin resistance is also a prominent component of cardiovascular diseases (CVD), including hypertension, coronary artery disease, and atherosclerosis, which are characterized by endothelial dysfunction. Insulin stimulates two distinct signaling pathways in the endothelium. One produces the vasodilator nitric oxide (NO) through the insulin receptor substrate-1(IRS-1)/endothelial NO synthase (eNOS) pathway while the other stimulates production of endothelin-1 (ET-1), a vasoconstrictor, through the mitogen activated protein kinase (MAPK) pathway. Insulin-mediated glucose disposal is largely dependent upon the vasodilatory effects of insulin; however, in T2D, insulin-stimulated dilation is impaired as a result of an imbalance in NO and ET-1 production, leading to diminished microvascular perfusion and skeletal muscle glucose delivery in response to insulin. The effects of exercise on insulin signaling/action in the endothelium are not fully understood. The purpose of this study is determine the acute effects of aerobic exercise training on cardiometabolic responses to meal ingestion in individuals with insulin resistance or T2D. We will recruit 30 previously sedentary (<60 minutes of planned exercise/week) men and women with insulin resistance (pre-diabetes) or T2D for participation in this study. Participants will undergo a screening procedure, including telephone screening and physical examination, as well as determination of body composition and fitness. Participants will be asked to complete 5-10 days of supervised exercise training and will undergo testing to assess cardiovascular and metabolic responses to an oral glucose tolerance test, including muscle sympathetic nerve activity, blood flow, and circulating glucose and insulin concentrations at baseline and following training. In addition, participants will use continuous glucose monitoring systems for 3 days at baseline and during 3 days of exercise training to assess the effects of acute exercise on postprandial glucose responses to mixed meals in free-living individuals. The overall aim of the project is to determine whether or not acute exercise training influences postprandial metabolic, vascular or autonomic nervous system responses in individuals with insulin resistance or T2D.

ELIGIBILITY:
Inclusion Criteria:

* Insulin resistant: diagnosed with pre-diabetes or fasting blood glucose >/= 100 mg/dL
* T2D: diagnosed by primary care physician
* BMI: less than 43 kg/m2
* Age: 30-65

Exclusion Criteria:

* Smoking
* Insulin use (other than once daily)
* Underlying conditions that limit ability to exercise safely
* Recent weight gain or loss (> 5% of body weight in 3 months)
* Physically active (> 30 min aerobic exercise, 2 d/wk)
* Recent (< 3 mo) changes in medication use or dose
* Uncontrolled T2D (HbA1c > 10%)
* Advanced retinopathy or neuropathy
* Pregnancy

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The overall aim of the project is to determine whether or not acute exercise training influences postprandial metabolic, vascular or autonomic nervous system responses in individuals with insulin resistance or T2D. | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: John P Thyfault, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Mikus CR, Oberlin DJ, Libla J, Boyle LJ, Thyfault JP. Glycaemic control is improved by 7 days of aerobic exercise training in patients with type 2 diabetes. Diabetologia. 2012 May;55(5):1417-23. doi: 10.1007/s00125-012-2490-8. Epub 2012 Feb 4. PMID 22311420
- [Derived] Mikus CR, Fairfax ST, Libla JL, Boyle LJ, Vianna LC, Oberlin DJ, Uptergrove GM, Deo SH, Kim A, Kanaley JA, Fadel PJ, Thyfault JP. Seven days of aerobic exercise training improves conduit artery blood flow following glucose ingestion in patients with type 2 diabetes. J Appl Physiol (1985). 2011 Sep;111(3):657-64. doi: 10.1152/japplphysiol.00489.2011. Epub 2011 Jul 7. PMID 21737826